CLINICAL TRIAL: NCT00972140
Title: A 3-month, Double-blind, Double-dummy, Randomised, Multinational, Multicenter, 2-arm Parallel-group Study Comparing the Efficacy and Safety of Formoterol-HFA pMDI 12µg Twice Daily and Formoterol-DPI 12µg Twice Daily, in Patients With Stable Chronic Obstructive Pulmonary Disease
Brief Title: Formoterol-HFA 3-month Study in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RA-PR-3301-011-04
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Patients with stable COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Formoterol-HFA (Experimental): Formoterol-HFA pMDI 12µg twice daily
  Interventions: Drug: Formoterol
- Formoterol-DPI (Active Comparator): Formoterol-DPI 12µg twice daily
  Interventions: Drug: Formoterol

INTERVENTIONS:
Drug: Formoterol — Formoterol-HFA pMDI 12µg twice daily
  Other Names: Atimos
  Arms: Formoterol-HFA
Drug: Formoterol — Formoterol-DPI 12 µg twice daily
  Other Names: Foradil
  Arms: Formoterol-DPI

SUMMARY:
The purpose of this study is to demonstrate the clinical equivalence of formoterol-HFA pMDI 12µg/actuation administered twice daily to formoterol DPI 12µg/capsule delivered by the Aerolizer inhaler and administered twice daily in patients with COPD.

DETAILED DESCRIPTION:
Phase III, multicenter, multinational, double-blind, double-dummy, randomised, 2-arm parallel-group, 3-month study in patients with stable COPD.

Comparison in terms of efficacy and safety of the two formulations of formoterol administered as 24µg/day in a bid regimen

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients who gave written informed consent.
* Diagnosis of stable COPD according to the recommendations of the -Diagnosis of stable COPD according to the recommendations of the National Heart Lung and Blood Institute (NHLBI) Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria, Edition 2003
* Age 40 years or older. Male and female patients who gave written informed consent
* History of a progressive nature of symptoms and a complaint of dyspnoea at least on exertion.
* Current or previous smoker [in both cases with a cumulative exposure to cigarette smoke of more than 20 pack-years
* Pre-bronchodilator baseline 40% > FEV1 < 70% of the predicted normal value
* Absolute value FEV1 > 0.9 L.
* FEV1/FVC < 70% (ERS criteria for predicted normal value).
* FEV1 reversibility test 30 minutes following inhalation of 400 μg of salbutamol pMDI
* A cooperative attitude and ability to be trained to use correctly the pMDI and the Aerolizer® inhaler

Exclusion Criteria:

* Female subjects: pregnant, lactating mother or lack of efficient contraception in a subject with childbearing potential (e.g. contraceptive methods other than oral contraceptives, IUD, tubal ligature).
* Current or past diagnosis of asthma.
* History of allergic rhinitis or other atopic disease (e.g. eczema).
* Largely reversible airflow obstruction.
* Onset of obstructive symptoms early in life (i.e. childhood).
* Variability of symptoms from day to day and frequent symptoms at night and early morning.
* A total blood eosinophil count higher than 500/μL.
* Significant and unstable concomitant cardiovascular, renal, hepatic, gastrointestinal,neurological, endocrine, metabolic, musculo-skeletal, neoplastic, respiratory or other clinically significant disease
* Clinical significant laboratory abnormalities indicating a significant or unstable concomitant disease.
* QTc interval (Bazett formula) higher than 460 msec
* Total 24 hours respiratory symptom score (day-time and night-time) > 2 on at least 4 consecutive days
* Lower respiratory tract infection within one month before screening visit
* Hospitalisation or emergency room treatment for an acute COPD exacerbation in the month before screening visit
* Long-term oxygen therapy.
* Patients treated with oral or injectable corticosteroids and antibiotics for a COPD exacerbation and/or a lower respiratory tract infection in the month preceding the screening visit and during the run-in period of the study.
* Patients treated with depot corticosteroids in the three months preceding the screening visit and during the 14-week study period.
* Changes in dose, schedule, formulation or product of an inhaled or nasal corticosteroid and oral modified-release theophylline within one month of screening visit and during the 14 week study period
* Patients treated with inhaled long-acting β2-agonists during the 14-week study period.
* Short-acting β2-agonists on regular use during the 14-week study period 8 hours preceding the screening visit
* Short-acting anticholinergic medications during the 14-week study period
* Long-acting anticholinergic medications (e.g. tiotropium) during the 14-week study period.
* Inhaled fixed combinations of a short-acting β2-agonist and a short-acting anticholinergic medication (e.g. Combivent) during the 14-week study period
* Inhaled fixed combinations of an inhaled corticosteroid and a long-acting β2-agonist (e.g.Seretide, Symbicort) during the 14-week study period.
* Long-acting antihistamines (e.g. Astemizole, Terfenadine) in the three months preceding the screening visit and during the 14-week study period.
* Tricyclic antidepressants, monoamine oxidase inhibitors (MAOI) and other drugs known to prolong the QTc interval during the 14-week study period.
* β-blockers in the week preceding the screening visit and during the 14-week study period.
* Intolerance to inhaled β2-adrenergic agents.
* History of intolerance or allergic reactions to any of the pMDI and DPI excipients.
* Patients who had evidence of alcohol or substance abuse, not compliant with the study protocol or not compliant with the study treatments.
* Participation in another clinical trial with an investigational drug in the four weeks preceding the screening visit

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2005-08; Primary Completion 2006-04 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
12-hour post-morning dose average FEV1 (area under the FEV1 versus time curve divided by 12 hours) after 12 weeks of treatment | Every 6 weeks

SECONDARY OUTCOMES:
Pulmonary Function tests :FEV1, FVC, symptom scores, COPD exacerbations, used of rescue | Every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Iwona Graelewska Rzymowska, Prof, Principal Investigator — Clinic Pneumology and Allergology Lodz Poland
Locations (1):
- Prof. Iwona Graelewska Rzymowska, Lodz, Lódz, Poland